CLINICAL TRIAL: NCT04628741
Title: Beyond the Dynamic Coaching Model: A Treatment Comparison for Undergraduate College Students With Traumatic Brain Injury
Brief Title: Treatment Comparison for Undergraduate College Students With Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 2010102285
Record Dates: First submitted 2020-10-05; First posted 2020-11-13 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Traumatic Brain Injury; Concussion, Brain
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Coaching Model (Active Comparator): The Dynamic Coaching Model is an established treatment approach that entails training college students with executive function impairments (e.g., those with a history of traumatic brain injury) to rely on their own executive functions in order to problem solve and reason in real-life situations requiring them to do so (e.g., taking college classes).
  Interventions: Behavioral: Dynamic Coaching Model
- Apprenticeship Approach for College Students (Experimental): The Apprenticeship Approach is a novel treatment approach that incorporates explicit education about: (a) traumatic brain injury definition; (b) traumatic brain injury symptomatology; and (c) individuals who may be able to provide assistance to the individual with traumatic brain injury into the existing Dynamic Coaching Model.
  Interventions: Behavioral: Apprenticeship Approach

INTERVENTIONS:
Behavioral: Dynamic Coaching Model — This is a behavioral intervention which includes metacognitive strategy training and personalized strategy and external aid use training.
  Arms: Dynamic Coaching Model
Behavioral: Apprenticeship Approach — This is a behavioral intervention which includes explicit education about traumatic brain injury, its symptoms, and individuals who may provide assistance post-injury, metacognitive strategy training and personalized strategy and external aid use training.
  Arms: Apprenticeship Approach for College Students

SUMMARY:
Up to 28% of undergraduate college students report a suspected history of traumatic brain injury. Following traumatic brain injury, college students fail and repeat more courses and have lower grade point averages. Further complicating this problem may be the fact that college students lack knowledge of traumatic brain injury definition, its associated symptoms, and individuals involved in post-injury management. In this project, the investigators propose to compare the use of an established treatment model (i.e., the Dynamic Coaching Model) to a novel protocol (i.e., the Apprenticeship Approach) that includes explicit instruction about traumatic brain injury in college students with this population. The investigators will use a group comparison design to examine the efficacy of this instructional component. This work incorporates findings from educational psychology and speech-language pathology (e.g., the included instructional materials adhere to the principles of adult learning). As such, this work will advance the field's basic understanding of currently recommended treatment components and will systematically examine the effects of incorporating explicit instruction into an existing treatment model.

ELIGIBILITY:
Inclusion Criteria:

* a documented history of mild, moderate, or severe traumatic brain injury no more than 36 months prior to study initiation
* speak English as a primary language
* at least 18 years of age
* demonstrate no barriers related to hearing, vision, reading, or technology that prevent successful experimental task completion.

Exclusion Criteria:

* no documented history of mild, moderate, or severe traumatic brain injury
* injury occurred more than 36 months prior to study initiation
* do not speak English as a primary language
* are not at least 18 years of age
* demonstrate barriers related to hearing, vision, reading, or technology that prevent successful experimental task completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Change in performance on a knowledge questionnaire | Up to 6 months (conducted once pre-intervention and once post-intervention)
  adapted from Knollman-Porter et al., 2017
Change in performance on measures of academic achievement | Up to 6 months (conducted once pre-intervention and once post-intervention)
  Self-Efficacy Scale (5-point scale)
Change in performance on measures of academic achievement | Up to 6 months (conducted once pre-intervention and once post-intervention)
  Self-Compassion Scale Short Form (5-point scale)
Change in performance on measures of academic achievement | 2 minutes (conducted once pre-intervention and once post-intervention)
  Growth Mindset Scale (5-point scale)
Change in performance on subjective confidence rankings | Up to 6 months (conducted once pre-intervention and once post-intervention)
  Confidence rankings on a 5-point Likert scale for therapy task performance and functional academic task performance
Performance on subjective intervention satisfaction rankings | Up to 6 months (conducted one time in each intervention session; i.e., three times total)
  Subjective rankings on a 5-point Likert scale for intervention satisfaction, likelihood to recommend intervention to a friend, and desire to continue intervention.
Change in performance on a measure of quality of life: QOLIBRI (Quality of Life After Brain Injury) | Up to 6 months (conducted once pre-intervention and once post-intervention)
  QOLIBRI (Quality of Life After Brain Injury)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States